CLINICAL TRIAL: NCT01170208
Title: Open-Label, Uncontrolled, Single-Arm, Single-Center, 16-Week Study Assessing Efficacy and Safety of Frequently Modified Insulin Therapy Using Dosage Recommending Device Software in 3-Groups of Subjects With Diabetes
Brief Title: Insulin Dosage Software Program for People With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Hygieia, Inc (Industry); International Diabetes Center at Park Nicollet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03985-10-A; R41DK085974 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-07-27 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2014-01

CONDITIONS: Diabetes; Insulin
Keywords: insulin; dosage software
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I (Other): Type 1 diabetes treated with basal-bolus insulin therapy, incorporating carbohydrate-counting and insulin dose software.
  Interventions: Device: insulin dose software
- Group II (Other): Type 2 diabetes treated with basal-bolustherapy and insulin dose software.
  Interventions: Device: insulin dose software
- Group III (Other): Type 2 diabetes treated with biphasic insulin and insulin dose software.
  Interventions: Device: insulin dose software

INTERVENTIONS:
Device: insulin dose software — The rationale to conduct this study is that Hygieia hypothesizes the software will effectively and safely optimize glucose control in insulin-requiring patients with type-1 and type-2 diabetes. The software was designed to provide safe insulin dosage recommendations.
  Other Names: blood glucose meter

SUMMARY:
The purpose of the study is to determine the effectiveness and safety of the computer software program in providing insulin dosage recommendations. Participation in the study for 60 research subjects will last for 16-weeks and includes 3-4 clinic visits and a series of weekly telephone calls from the study team (minimum of 12 calls). Participants will be provided with weekly Study Log Sheets to record their daily blood glucose readings, insulin doses, grams of carbohydrate eaten at each meal (if they have type-1 diabetes) and any changes in their health (e.g., hypoglycemic episodes, illnesses). Participants will fax or drop off a copy of the Study Log Sheet. This information will be entered by the IDC study team into the computer software program. The IDC study team will review the information from the software and, based on the IDC's study team approval, any insulin dose changes will be communicated back to the patient by phone or fax.

DETAILED DESCRIPTION:
Hygieia, Inc. is developing a device intended for use by insulin-requiring patients with diabetes. It will be a pocket-sized, hand-held device, combining a glucose meter with software that analyzes blood glucose levels recorded in the device's memory, and periodically recommends modifications in insulin dosage. The already developed software algorithms are based on the way an endocrinologist evaluates and frequently adjusts insulin dosage in a patient with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* GROUP I
* Have been clinically diagnosed with type-1 diabetes for at least 1-year
* Have an HgbA1c of 7.4% or higher
* Treated with short-acting insulin analog (i.e. HumaLog® Lispro, NovoLog® Aspart, Apidra® Glulisine) before each meal and only one injection of long-acting insulin analog Lantus® (Glargine), per day. Subjects must typically eat 3 meals per day. The total daily combined dose of the long-acting and short-acting insulin analogs must be 25 units or more. Patient must have been using the same insulin regimen for the previous 3-months
* Is currently using an insulin/carbohydrate ratio to decide how much short-acting insulin to take before meals and must be able to use the gram versus choice method of carbohydrate counting.
* GROUP II
* Have been clinically diagnosed with type-2 diabetes for at least 1-year
* Have an HgbA1c of 7.4% or higher
* Treated with short-acting insulin analog (i.e. HumaLog® Lispro, NovoLog® Aspart, Apidra® Glulisine) before each meal and only one injection of long-acting insulin analog Lantus® (Glargine) per day and. Subjects must typically eat 3 meals per day. The total daily combined dose of the long-acting and short-acting insulin analogs must be 25 units or more. Patient must have been using the same insulin regimen for the previous 3-months
* May be using other diabetes agent(s) at a stable dose for the last 3-months.
* GROUP III
* Have been clinically diagnosed with type-2 diabetes for at least 1-year
* Have an HgbA1c of 7.8% or higher
* Take twice daily biphasic Insulin (e.g. HumaLog® Mix 75/25, NovoLog® Mix 70/30) or premixed insulin (i.e. Humulin® 70/30, Novolin® 70/30, NPH/Regular insulin 70/30) with a total daily insulin dose of 25 units and have been using the same insulin regimen for the past 3-months
* May be using other diabetes agent(s) at a stable dose for the last 3-months.

Exclusion Criteria:

* Have a history of greater than 2 episodes of severe hypoglycemia in the past year, or have hypoglycemic unawareness when glucose levels are less than or equal to 50 mg/dl
* Have a significant physical, psychological, or cognitive impairment that would prohibit adherence to the protocol
* Have any severe cardiovascular disease including a history of congestive heart failure (New York Heart Association [NYHA] 3 or 4), unstable angina, myocardial infarction or stroke that occurred within the 6-months preceding enrollment
* Have known active anemia with a hemotocrit less than 25% in women or 30% in men
* Have known history of renal disease (e.g., serum creatinine level >2.0 mg/dl or eGFR < 30 ml/min)
* Have active cancer or cancer in the past 2-years (except non-melanoma skin cancer
* Have history of significant liver disease including cirrhosis or elevated liver enzymes (e.g., AST and ALT greater than 3 times the upper limit of normal values)
* Have a body mass index (BMI) > 45 kg/m2; and/or
* Are pregnant, plan to become pregnant during the study period, or are breastfeeding.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bergenstal, MD, Principal Investigator — International Diabetes Center at Park Nicollet; Eran Bashan, PhD, Study Director — Hygieia, Inc
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Herman WH, Ilag LL, Johnson SL, Martin CL, Sinding J, Al Harthi A, Plunkett CD, LaPorte FB, Burke R, Brown MB, Halter JB, Raskin P. A clinical trial of continuous subcutaneous insulin infusion versus multiple daily injections in older adults with type 2 diabetes. Diabetes Care. 2005 Jul;28(7):1568-73. doi: 10.2337/diacare.28.7.1568. PMID 15983302
- [Background] Bergenstal RM, Johnson M, Powers MA, Wynne A, Vlajnic A, Hollander P, Rendell M. Adjust to target in type 2 diabetes: comparison of a simple algorithm with carbohydrate counting for adjustment of mealtime insulin glulisine. Diabetes Care. 2008 Jul;31(7):1305-10. doi: 10.2337/dc07-2137. Epub 2008 Mar 25. PMID 18364392
- [Derived] Bergenstal RM, Bashan E, McShane M, Johnson M, Hodish I. Can a tool that automates insulin titration be a key to diabetes management? Diabetes Technol Ther. 2012 Aug;14(8):675-82. doi: 10.1089/dia.2011.0303. Epub 2012 May 8. PMID 22568777
- See also: Publication — http://www.ncbi.nlm.nih.gov/pubmed/22568777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2010 to October 2010. Location: Medical Clinic
Groups:
- Group I: Type 1 diabetes treated with basal-bolus insulin therapy, incorporating carbohydrate-counting
- Group II: Type 2 diabetes treated with basalbolus therapy
- Group III: Type 2 diabetes treated with biphasic insulin.
Period: Overall Study
Arm/Group | Group I | Group II | Group III
Started | 20 | 20 | 6
Completed | 14 | 20 | 4
Not Completed | 6 | 0 | 2
Not completed — Withdrawal by Subject | 5 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Group III | Total
Number analyzed (Participants) | 20 | 20 | 6 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 13 | 5 | 38
  >=65 years | 0 | 7 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12) | 60 (7) | 55 (7) | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 4 | 27
  Male | 7 | 10 | 2 | 19
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 6 | 46
Weekly Mean Blood Glucose [Mean (Standard Deviation); unit: mg/dL] — Week 4 baseline weekly mean blood glucose
  mg/dL | 176.9 (28.3) | 164.9 (37.6) | 190.8 (47.0) | 172.4 (35.0)
HbA1c [Mean (Standard Deviation); unit: percent] | 8.4 (0.6) | 8.3 (0.8) | 9.1 (1.5) | 8.4 (0.8)
Fructosamine [Mean (Standard Deviation); unit: µM] | 349 (46) | 273 (30) | 270 (33) | 303 (53)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Mean Blood Glucose From Week 4 to Week 16
Time Frame: Twelve week period from week 4 to week 16
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Group I: Type 1 diabetes treated with basal-bolus insulin the
- Group II: Type 2 diabetes treated with basal bolus therapy
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 14 | 20 | 4
mg/dL | 4.6 (29.3) | 8.1 (51.0) | 29.5 (17.1)

2. Secondary Outcome: Reduction in HbA1c.
Time Frame: Twelve week period from week 4 to week 16
Measure: Mean (Standard Deviation); unit: percentage of A1c
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 20 | 20 | 6
percentage of A1c | 0.1 (0.8) | 0.6 (0.9) | 1.3 (1.4)

3. Secondary Outcome: Reduction in Fructosamine.
Time Frame: 12 week period from Week 4 to Week 16
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 20 | 20 | 6
µM | -4.2 (29.2) | 10.2 (32.2) | 37.0 (20.9)

4. Secondary Outcome: Incidence of Severe or Serious Hypoglycemia.
Time Frame: January 2011
Measure: Count of Participants; unit: Participants
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 20 | 20 | 6
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group I | Group II | Group III
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/6
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/6

LIMITATIONS AND CAVEATS:
Study was limited by lack of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes